CLINICAL TRIAL: NCT06767917
Title: Safety and Performance of the Ophthalmic Viscoelastic Devices Eyefill SC and Eyefill MB - a Post-Market Clinical Follow-Up
Brief Title: A Post-Market Clinical Follow-Up on Safety and Performance of the Ophthalmic Viscoelastic Devices Eyefill SC and Eyefill MB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb GmbH (Industry)
Responsible Party: Sponsor
Organization: Bausch & Lomb Incorporated (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 931
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eyefill® S.C. (Experimental)
  Interventions: Device: Eyefill® S.C.
- Eyefill® M.B. (Experimental)
  Interventions: Device: Eyefill® M.B.

INTERVENTIONS:
Device: Eyefill® S.C. — Used as viscoelastic devices during cataract surgery
  Arms: Eyefill® S.C.
Device: Eyefill® M.B. — Used as viscoelastic devices during cataract surgery
  Arms: Eyefill® M.B.

SUMMARY:
Prospective, Non-comparative, Post Market Clinical Follow Up Study to demonstrate safety and performance of Eyefill® S.C. and Eyefill® M.B. as viscoelastic devices for cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects scheduled for cataract surgery with im-plantation of a posterior chamber intraocular lens;
* Signed informed consent;
* Availability, willingness, ability, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Known hypersensitivity to sodium hyaluronate;
* Corneal endothelial cell density <1500 cells/mm2;
* Corneal abnormalities;
* Cataract density of grade 4+;
* Previous intraocular or corneal surgery;
* Chronic or recurrent inflammatory eye diseases (e.g., iritis, scleritis, iridocyclitis, or rubeosis iridis);
* Clinically significant, uncontrolled glaucoma with expected negative impact on visual acuity outcomes;
* Ongoing systemic or ocular steroid therapy;
* Diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity loss to 20/30 or worse in one or both eyes;
* Active ocular or systemic infection (bacterial, viral, or fungal), including fever
* Subjects who may be expected to require a combined or other secondary surgical procedure
* Females of childbearing potential (those who are not surgically sterilized or not postmenopausal for at least 12 months) if they meet one of the following conditions: Pregnant, lactating or unwilling to use effective birth control over the course of the study;
* Concurrent or previous (within 30 days) participation in another drug or device investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in corneal endothelial cell density between baseline and postoperative visits | Assessed on Day 30 and Day 90

OTHER OUTCOMES:
Safety outcome - Adverse event rate | Assessed up to Day 90

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Site 102, Madrid
  - Site 103, Zaragoza

IPD SHARING:
Plan to Share IPD: No